CLINICAL TRIAL: NCT00301457
Title: A Prospective Randomised, Open, Multicentre, Phase III Study to Assess Different Durations of Anastrozole Therapy After 2 to 3 Years Tamoxifen as Adjuvant Therapy in Postmenopausal Women With Breast Cancer.
Brief Title: Different Durations of Adjuvant Anastrozole Therapy After 2 to 3 Years Tamoxifen Therapy in Breast Cancer
Acronym: DATA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5392NL003; EUDRAct No: 2005-006167-31
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Hormone Sensitive Primary Breast Cancer; Adjuvant Treatment; Aromatase Inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

ARMS (2):
- 1 (Experimental): 6 years adjuvant anastrozole therapy
  Interventions: Drug: Anastrozole
- 2 (Experimental): 3 years adjuvant anastrozole therapy
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1 mg once daily oral dose
  Other Names: ARIMIDEX; ZD1033

SUMMARY:
The purpose of this study is to determine whether 6 years adjuvant anastrozole will improve the disease free survival compared to 3 years adjuvant anastrozole in postmenopausal hormone sensitive breast cancer patients, subsequent to 2-3 years tamoxifen

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal patients with hormone receptor positive breast cancer who have already received 2 to 3 years of adjuvant tamoxifen, and who never had signs of loco-regional recurrences or distant metastasis

Exclusion Criteria:

* Previous hormonal therapy as adjuvant breast cancer treatment besides tamoxifen.
* Previous history of invasive breast cancer within the last 10 years, other then the breast cancer that is currently treated with tamoxifen

Ages: 45 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1914 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
To assess the disease free survival (DFS) with 6 years of adjuvant anastrozole compared with 3 years of adjuvant anastrozole in postmenopausal hormone sensitive breast cancer patients, subsequent to 2 to 3 years of adjuvant tamoxifen | After 9 years for the group with 6 years of adjuvant anastrozol, subsequent to 2 to 3 years of adjuvant tamoxifen or after 6 years for the group with 3 years of adjuvant anastrozole subsequent to 2 to 3 years of adjuvant tamoxifen

SECONDARY OUTCOMES:
To compare the incidence of contralateral breast cancer after 6 years versus 3 years adjuvant anastrozole, subsequent to 2 to 3 years of tamoxifen | After 9 years for the group with 6 years of adjuvant anastrozol, subsequent to 2 to 3 years of adjuvant tamoxifen or after 6 years for the group with 3 years of adjuvant anastrozole subsequent to 2 to 3 years of adjuvant tamoxifen
To compare the overall survival after 6 years versus 3 years adjuvant anastrozole, subsequent to 2 to 3 years of tamoxifen | After 9 years for the group with 6 years of adjuvant anastrozol, subsequent to 2 to 3 years of adjuvant tamoxifen or after 6 years for the group with 3 years of adjuvant anastrozole subsequent to 2 to 3 years of adjuvant tamoxifen
To compare toxicity of 6 years versus 3 years of adjuvant anastrozole in postmenopausal hormone sensitive breast cancer patients, subsequent to 2 to 3 years of tamoxifen | After 9 years for the group with 6 years of adjuvant anastrozol, subsequent to 2 to 3 years of adjuvant tamoxifen or after 6 years for the group with 3 years of adjuvant anastrozole subsequent to 2 to 3 years of adjuvant tamoxifen
To determine regional differences in the initial treatment of breast cancer retrospectively by collecting baseline information on initial therapies. | After 9 years
  Aspects of the initial treatment that will be investigated are e.g. the kind of surgery performed (breast saving or mastectomy) and whether or not chemotherapy is given and which chemotherapy was used in postmenopausal patients in relation to the primary tumour and patient characteristics.
To compare the cost effectiveness of 3 years versus 6 years adjuvant anastrozole therapy, after subsequent 2 to 3 years of adjuvant tamoxifen treatment. | After 9 years for the group with 6 years of adjuvant anastrozol, subsequent to 2 to 3 years of adjuvant tamoxifen or after 6 years for the group with 3 years of adjuvant anastrozole subsequent to 2 to 3 years of adjuvant tamoxifen
To assess patterns of care in The Netherlands in prevention, detection and treatment of osteoporosis in postmenopausal women with breast cancer treated with adjuvant anastrozole. | After 9 years
To relate the number of osteoporotic fractures during and following treatment with adjuvant anastrozole with the compliance to osteoporotic guidelines. | After 9 years
To analyse occurrence of distant (bone) metastases in relation to occurrence of osteopenia and osteoporosis, and in relation to use of supplements and therapy for reduced BMD. | After 9 years

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (67):
- Netherlands (67):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Almere Stad
  - Research Site, Amersfoort
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Arnhem
  - Research Site, Bergen op Zoom
  - Research Site, Beugen
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Deventer
  - Research Site, Dirksland
  - Research Site, Doetinchem
  - Research Site, Dordrecht
  - Research Site, Drachten
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Emmen
  - Research Site, Enschede
  - Research Site, Flushing
  - Research Site, Geldrop
  - Research Site, Geleen
  - Research Site, Goes
  - Research Site, Gorinchem
  - Research Site, Gouda
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Hengelo
  - Research Site, Hilversum
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Leeuwarden
  - Research Site, Leiden
  - Research Site, Leidschendam
  - Research Site, Maastricht
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Purmerend
  - Research Site, Roermond
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Sneek
  - Research Site, Spijkenisse
  - Research Site, Stadskanaal
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Uden
  - Research Site, Utrecht
  - Research Site, Veldhoven
  - Research Site, Venlo
  - Research Site, Winschoten
  - Research Site, Winterswijk
  - Research Site, Woerden
  - Research Site, Zaandam
  - Research Site, Zevenaar
  - Research Site, Zoetermeer
  - Research Site, Zutphen
  - Research Site, Zwolle

REFERENCES:
- [Derived] Tjan-Heijnen VCG, Lammers SWM, Geurts SME, Vriens IJH, Swinkels ACP, Smorenburg CH, van der Sangen MJC, Kroep JR, de Graaf H, Honkoop AH, Erdkamp FLG, de Roos WK, Linn SC, Imholz ALT; Dutch Breast Cancer Research Group (BOOG) for the DATA Investigators. Extended adjuvant aromatase inhibition after sequential endocrine therapy in postmenopausal women with breast cancer: follow-up analysis of the randomised phase 3 DATA trial. EClinicalMedicine. 2023 Mar 20;58:101901. doi: 10.1016/j.eclinm.2023.101901. eCollection 2023 Apr. PMID 36992863
- [Derived] van Hellemond IEG, Smorenburg CH, Peer PGM, Swinkels ACP, Seynaeve CM, van der Sangen MJC, Kroep JR, de Graaf H, Honkoop AH, Erdkamp FLG, van den Berkmortel FWPJ, de Boer M, de Roos WK, Linn SC, Imholz ALT, Tjan-Heijnen VCG; Dutch Breast Cancer Research Group (BOOG). Assessment and management of bone health in women with early breast cancer receiving endocrine treatment in the DATA study. Int J Cancer. 2019 Sep 1;145(5):1325-1333. doi: 10.1002/ijc.32205. Epub 2019 Mar 4. PMID 30748011
- [Derived] van Hellemond IEG, Vriens IJH, Peer PGM, Swinkels ACP, Smorenburg CH, Seynaeve CM, van der Sangen MJC, Kroep JR, de Graaf H, Honkoop AH, Erdkamp FLG, van den Berkmortel FWPJ, de Boer M, de Roos WK, Linn SC, Imholz ALT, Tjan-Heijnen VCG; Dutch Breast Cancer Research Group (BOOG). Efficacy of anastrozole after tamoxifen in early breast cancer patients with chemotherapy-induced ovarian function failure. Int J Cancer. 2019 Jul 1;145(1):274-283. doi: 10.1002/ijc.32093. Epub 2019 Jan 16. PMID 30588619
- [Derived] Tjan-Heijnen VCG, van Hellemond IEG, Peer PGM, Swinkels ACP, Smorenburg CH, van der Sangen MJC, Kroep JR, De Graaf H, Honkoop AH, Erdkamp FLG, van den Berkmortel FWPJ, de Boer M, de Roos WK, Linn SC, Imholz ALT, Seynaeve CM; Dutch Breast Cancer Research Group (BOOG) for the DATA Investigators. Extended adjuvant aromatase inhibition after sequential endocrine therapy (DATA): a randomised, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1502-1511. doi: 10.1016/S1470-2045(17)30600-9. Epub 2017 Oct 12. PMID 29031778

DOCUMENTS (1):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT00301457/Prot_000.pdf